CLINICAL TRIAL: NCT01132599
Title: A Cancer Research UK Phase II Trial to Compare [11C]Choline and [18F]Choline Each Given as a Single Administration Via Intravenous Injection for Imaging Patients With Metastatic Prostate Cancer
Brief Title: Comparing PET-CT Using C-11 Choline and 18F-Fluoromethylcholine in Patients With Metastatic Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000674024; CRUK-CR0701-21; EUDRACT-2008-004828-23
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluoromethylcholine

INTERVENTIONS:
Dietary Supplement: C-11 choline
Radiation: 18F-fluoromethylcholine

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET) and computed tomography (CT) imaging, may help find and diagnose metastatic prostate cancer.

PURPOSE: This phase II trial is studying the side effects of C-11 choline and 18F-fluoromethylcholine and to see how well they work when used in PET and CT imaging in patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare C-11 choline to 18F-fluoromethylcholine using positron emission tomography and computed tomography imaging in their ability to detect metastatic prostate cancer.
* To compare the best early-phase (immediate) scanning of the two agents against the late-phase (one-hour delayed) 18F-fluoromethylcholine scanning in their ability to detect metastatic prostate cancer.
* To assess the safety of C-11 choline and 18F-fluoromethylcholine in these patients.

OUTLINE: Patients receive C-11 choline IV followed by a 10-minute dynamic positron emission tomography (PET) scan over the pelvis and then 5-minute scans at each bed position, from the pelvis to the base of the skull, (up to a maximum of 7 additional bed positions) lasting up to 45 minutes on day 1. Beginning 3 hours later, patients receive 18F-fluoromethylcholine IV followed by the same scanning protocol above lasting approximately 45 minutes. An additional 1-hour delayed PET-computed tomography (CT) scanning is then performed, which involves a 5-minute scan at each bed position from the pelvis to the base of the skull (up to a maximum of 7 bed positions) with 18F-fluoromethylcholine, lasting approximately 35 minutes. Patients then undergo treatment as per the normal standard of care following participation in this trial.

After completion of study treatment, patients are followed between 3-7 days.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* At least 4 metastatic lesions identified by conventional imaging with bone scintigraphy
* Treatment-naive disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN if due to tumor)
* Fertile patients must use two forms of effective contraception 2 weeks prior to, during, and for 6 months after completion of study therapy
* None of the following conditions that would prevent compliance with the study protocol:

  * Diabetes
  * High levels of pain/discomfort
  * Urinary incontinence
* No history of recent significant cardiac arrhythmia
* No concurrent congestive heart failure or prior history of NYHA class III-IV cardiac disease
* No other condition that, in the investigator's opinion, would not make the patient a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy, hormone therapy, chemotherapy, endocrine therapy, or immunotherapy for the treatment of prostate cancer
* No major thoracic and/or abdominal surgery from which the patient has not yet recovered
* No concurrent anticancer therapy
* No concurrent hormone therapy
* No concurrent participation or planning to participate in another interventional clinical trial

  * Concurrent participation in an observational trial allowed
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Identification of a true 5% difference in lesion detection using 18F-fluoromethylcholine versus C-11 choline

SECONDARY OUTCOMES:
Identification of a true 5% difference in lesion detection between the best early-phase scanning, using either the 18F-fluoromethylcholine and C-11 choline, and late-phase scanning using 18F-fluoromethylcholine
Causality of each adverse event to C-11 choline and 18F-fluoromethylcholine and adverse event severity according to NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Doherty, MD, Principal Investigator — St. Thomas' Hospital
Locations (1):
- St. Thomas' Hospital, London, England, United Kingdom